CLINICAL TRIAL: NCT01758419
Title: The Role of Myocardial SPECT in Evaluation of Irradiation-induced Changes With Myocardial Perfusion, Cardiac Function, Metabolism and Clinical Prognosis.
Brief Title: The Role of Myocardial SPECT in Evaluation of Irradiation-induced Changes.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-IRB-101085-F
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer, Female
Keywords: post-RT; myocardial perfusion images
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood sampling
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tomotherapy: Breast cancer female s/p scheduled RT will be arranged to undergo Thallium-201 Myocardial Perfusion Study. The scheduled RT will be arranged by clinical judgments of radiation-oncologists. All of the patients will receive myocardial SPECT before and after the scheduled RT. Comparing the clinical follow-up data between different groups (left-sided s/p tomography, left-sided s/p conventional RT, and right-sided RT), respectively.
  Interventions: Radiation: Thallium-201 Myocardial Perfusion Study

INTERVENTIONS:
Radiation: Thallium-201 Myocardial Perfusion Study — One-day Tl-201 stress/rest MPI protocol with pharmacological stress, as daily practice will be applied. CZT camera with multipinhole collimator and stationary detectors scan heart simultaneously. A 10% symmetrical energy window at 140 keV was used. Electrocardiogram-gated scans will be applied. Perfusion images were reconstructed in standard axis and polar maps of the left ventricle were obtained. Scans from CZT was analyzed in consensus by two experienced readers blinded to any information on patient identification. The software package Myovation for Alcyone, QGS and QPS were used for quantitative analysis of MPI polar maps. Automated analysis to determine ejection fraction.

SUMMARY:
Helical tomotherapy nowadays provides the most precise data on radiotherapy (RT) dose delivered to each region of the heart in left-sided breast cancer therapy, which allows greater sparing of the heart from doses associated with increased complications. However, heart disease shows a wide spectrum of pathologies, and multiple risk factors related. The damage of the myocytes may lead to not only myocardial perfusion defects, but also in functional deterioration, or even in biomarkers. In this study, we will monitor cardiovascular (CV) risk factors, metabolism, biomarkers, myocardial perfusion defect patterns, and cardiac functional parameters, in order to delineate of RT-related effects and clinical impacts.

Objective: The pilot study aims to investigate the correlation of post-tomotherapy cardiovascular effects with myocardial perfusion and cardiac functional studies.

Methods: The study plans to enroll female breast cancer patients who will undergo local RT after their surgery. Patients will receive global risk scoring assessment (Framingham Risk Score, FRS), blood sampling for basic biochemistry, inflammatory biomarker, and myocardial perfusion image (MPI) at the time points of before and after RT. The results of MPI will be analyzed in qualitative visual interpretation of perfusion patterns, and functional quantitative data for cardiac functional parameters as well. The patients will be regular followed-up in CV OPD. The association between baseline and follow-up MPI, biomarker and clinical presentation will be further investigated.

DETAILED DESCRIPTION:
* Inclusion Criteria:

  1. Female patients with breast cancer who scheduled further regional RT. Groups of left-sided breast cancer (tomotherapy, conventional RT), and right breast cancer (conventional RT).
  2. Aged 20-80 years old.
* Exclusion Criteria

  1. Pre-existing cardiac disease, such as prior myocardial infarction, documented CAD, congestive heart failure.
  2. Pregnancy
  3. Any medical contraindication of cardiac SPECT.
* Estimated Case Number 20 female patients of each groups, respectively Group 1: Left-sided breast cancer, planning to received helical tomography Group 2: Left-sided breast cancer, planning to received local conventional RT Group 3: Right-sided breast cancer, planning to received local RT

  1. Patients with breast cancer s/p operation will be transferred to CV OPD for initial cardiovascular risk factors assessment.
  2. Past history, family history, basic lab data and Framingham cardiovascular risk assessment will be applied. Intermediated to high risk need further work-up, and undergo SPECT before further RT course.
  3. All enrolled subjects provide basic demographic data and sign informed consents.
  4. Myocardial perfusion images for baseline evaluation before RT.
  5. The patients received scheduled treatment plan, including RT.
  6. Follow-up CV OPD every 3 months.
  7. Post-therapeutic myocardial perfusion study 12 months after first CV OPD visit.
  8. Comparing the clinical follow-up data between groups, including global functional assessments, blood sampling data, myocardial perfusion scan, and quantitative cardiac functional parameters.

Blood sampling

Myocardial perfusion study- Patients referred for SPECT MPI for evaluation of CAD underwent a 1-day Tl-201 stress/rest MPI protocol, as daily practice in FEMH. Pharmacological stress was induced by standard dipyridomale infusion. Tl-201 of 2 mCi was injected after 7 min of induced stress. Each scan will be performed on an ultrafast CZT camera (Discovery 530 NMc, GE Healthcare). CZT images were reconstructed on the workstation using a dedicated iterative algorithm with maximum likelihood expectation maximization. Perfusion images in standard axis (short axis, vertical long axis, horizontal long axis) and polar maps of the left ventricle were obtained. Scans from CZT was analyzed in consensus by two experienced readers blinded to any information on patient identification.

The software package with a 17-segment model for the left ventricle. Automated analysis of gated acquisitions from high-dose (rest) scans was performed to determine left ventricular ejection fraction. Integrated clinical information, follow-up and nuclear medicine cardiac scans performed in the time points of before & after RT will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer who scheduled further regional RT. Groups of left-sided breast cancer (tomotherapy, conventional RT), and right breast cancer (conventional RT).
* Aged 20-80 years old.

Exclusion Criteria:

* Pre-existing cardiac disease, such as prior myocardial infarction, documented CAD, congestive heart failure.
* Pregnancy
* Any medical contraindication of cardiac SPECT.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with breast cancer who scheduled further regional RT. Groups of left-sided breast cancer (tomotherapy, conventional RT), and right breast cancer (conventional RT).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
To investigate the correlation of post-RT cardiovascular effects with myocardial Tl-201 myocardial perfusion images | Dec, 2013 (after 12 months of baseline study).
  By literature reviewing, cardiovascular functional status in patients received helical tomography has not been fully investigated yet. And the post-therapeutic heart disease tends to show a wide spectrum of pathologies and multiple risk factors. We will monitor risk factors of underlying disease, family history, metabolism, biomarkers, myocardial perfusion defect patterns, and cardiac functional parameters, in order to delineation of RT-related effects and clinical prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Ying Wang, M.D., Principal Investigator — Far Eastern Memorial Hospital, Taiwan
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

REFERENCES:
- [Derived] Wang SY, Lin KH, Wu YW, Yu CW, Yang SY, Shueng PW, Hsu CX, Wu TH. Evaluation of the cardiac subvolume dose and myocardial perfusion in left breast cancer patients with postoperative radiotherapy: a prospective study. Sci Rep. 2023 Jun 29;13(1):10578. doi: 10.1038/s41598-023-37546-7. PMID 37386034